CLINICAL TRIAL: NCT00143325
Title: An Open-Label, Multicenter Study With Follow-Up Evaluating the Safety and Efficacy of Varenicline Tartrate in Comparison to Transdermal Nicotine Patch for Smoking Cessation
Brief Title: An Open Label Study That Compares Varenicline to Transdermal Nicotine Patch for Smoking Cessation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051044
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline (CP-526,555)

SUMMARY:
Open-label comparison of standard 12-week regimen of varenicline with standard 10-week regimen of transdermal nicotine patch for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have smoked an average of at least 15 cigarettes per day during the past year and over the month prior to the screening visit, with no period of abstinence greater than 3 months in the past year.

Exclusion Criteria:

* Subjects with clinically significant cardiovascular disease in the past 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730
Dates: Start 2005-01; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Continuous abstinence for the last 4 weeks of varenicline and NRT (Nicotine Replacement Therapy) treatment period

SECONDARY OUTCOMES:
Continuous abstinence last 4 weeks of treatment through Weeks 24 and 52
7-day point prevalence of abstinence: end of treatment, Weeks 24 and 52
4-week Point Prevalence of abstinence at Week 52
Long-Term Quit Rate at Weeks 24 and 52
Minnesota Nicotine Withdrawal Scale
Smoking Effects Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (6):
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Portland, Oregon
- Belgium (3):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
- France (6):
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Limeil-Brévannes
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Netherlands (4):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Enschede
  - Pfizer Investigational Site, Maastricht
  - Pfizer Investigational Site, Zutphen
- United Kingdom (3):
  - Pfizer Investigational Site, London, Surrey
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Nottingham

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Aubin HJ, Bobak A, Britton JR, Oncken C, Billing CB Jr, Gong J, Williams KE, Reeves KR. Varenicline versus transdermal nicotine patch for smoking cessation: results from a randomised open-label trial. Thorax. 2008 Aug;63(8):717-24. doi: 10.1136/thx.2007.090647. Epub 2008 Feb 8. PMID 18263663
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051044&StudyName=An+Open+Label+Study+that+Compares+Varenicline+to+Transdermal+Nicotine+Patch+for+Smoking+Cessation